CLINICAL TRIAL: NCT05777889
Title: The Effect of Spinal Cord Stimulation on Thermal Forward Looking InfraRed (FLIR) Imaging in Complex Regional Pain Syndrome (CRPS)
Brief Title: Infrared Images for Spinal Cord Stimulation in Complex Regional Pain Syndrome Patients
Acronym: SCS-FLIR
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2480
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Complex Regional Pain Syndromes
Keywords: spinal; infrared
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study CRPS Group: Enrolled patients with complex regional pain syndrome undergoing a surgical procedure that requires spinal cord stimulation.
  All participants in the group will have an image of their feet taken perpendicularly with a 1-inch space from all four sides using a FLIR T420 or T62101 camera with 320*240 resolution.
  All participants will also answer questionnaires about: their average pain score, CRPS severity, and neuropathic pain.
  Interventions: Other: Forward Looking InfraRed Camera

INTERVENTIONS:
Other: Forward Looking InfraRed Camera — Forward Looking InfraRed Camera:
  1. We will use a FLIR T420 or T62101 camera with a resolution of 320*240.
  2. Each image will be captured perpendicularly with a 1-inch gap on all four sides.
  3. A Myler blanket placed in the background will separate the feet from the background.
  4. The camera will be normalized to a temperature range of 15°C to 40°C.
  5. The images will be saved in radiometric JPEG format.
  6. Once the images have been transferred to a computer, we will remove the background.
  7. Next, we'll make a temperature histogram with 0.1°C temperature bin resolution.
  8. The before and after histograms (IB, IA) will be compared to see which one indicates more extreme temperature distributions.
  9. Those who improve by 30% or more are considered to have had a successful spinal cord stimulation.

SUMMARY:
The goal of this observational study is to compare thermal camera Forward Looking InfraRed (FLIR) images before and after spinal cord stimulation to evaluate the difference in sympathetic activity of the affected limb in patients with complex regional pain syndrome (CRPS). The main questions it aims to answer are:

Question 1: Can Infrared (FLIR) imaging be used to monitor the sympatholytic activity caused by Spinal Cord Stimulation (SCS) in patients with CRPS?

Question 2: Is there any correlation between the quantification of sympatholytic activity produced by Spinal Cord Stimulation (SCS) and measured by FLIR imaging with the outcome measures in patients with CRPS? Outcome measures include pain (NRS), CRPS Severity Score (CSS), and neuropathic pain score (painDETECT).

Participants will have an image of their feet taken perpendicularly with a 1-inch space from all four sides using a FLIR T420 or T62101 camera with 320*240 resolution.

Participants will also complete questionnaires about the average pain, CRPS severity, and neuropathic pain.

DETAILED DESCRIPTION:
Patients with CRPS often present with sympathetic dysfunction and peripheral vasomotor disturbances. Spinal Cord Stimulation (SCS) may have a sympatholytic effect with improved microcirculation and regional blood flow. This research proposal aims to investigate the potential use of Forward Looking Infrared (FLIR) imaging to monitor whether the sympatholytic effect is enhanced by using SCS in CRPS patients. The goal of this observational study is to compare thermal camera Forward Looking InfraRed (FLIR) images before and after spinal cord stimulation to evaluate the difference in sympathetic activity of the affected limb in patients with complex regional pain syndrome (CRPS). The main questions it aims to answer are:

Question 1: Can Infrared (FLIR) imaging be used to monitor the sympatholytic activity caused by Spinal Cord Stimulation (SCS) in patients with CRPS?

Question 2: Is there any correlation between the quantification of sympatholytic activity produced by Spinal Cord Stimulation (SCS) and measured by FLIR imaging with the outcome measures in patients with CRPS? Outcome measures include pain (NRS), CRPS Severity Score (CSS), and neuropathic pain score (painDETECT).

Participants will have an image of their feet taken perpendicularly with a 1-inch space from all four sides using a FLIR T420 or T62101 camera with 320*240 resolution.

Participants will also complete questionnaires about the average pain, CRPS severity, and neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* The patient is between 18 and 85 years old
* Providing CRPS diagnostic criteria by using the Budapest Clinical Diagnostic Criteria.
* CRPS affecting unilateral lower extremity
* The patient has had pain and other symptoms for more than 3 months
* Not responding to conventional medical treatments and multidisciplinary approach
* High NRS detection in pain assessment despite appropriate treatment (NRS= and > 6/10).
* Pain causing a limitation in the patient's functional capacity despite appropriate treatment.

Exclusion Criteria:

* Patients with suspected disc herniation, spinal stenosis, myelopathy, and suspected radiculopathy in detailed examinations and examinations (MRI, CT).
* Systemic or local infection
* Coagulation disorders
* History of allergy to contrast material
* Malignancy
* Pregnancy
* Uncontrollable medical and psychiatric condition
* The patients diagnosed with dysautonomia, sympathetic dysfunction other than CRPS (such as Raynaud disease or Buerger disease), sweating disorders other than CRPS (such as acquired idiopathic generalized anhidrosis), and patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosised with complex regional pain syndrome, undergoing a surgery that requires spinal cord stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Temperature difference in limb | 2-8 days after the trial procedure
  The temperature of the limb will be measured using the forward-looking infrared camera. A 30% or more improvement in temperature difference in the affected limb 2-8 days after spinal cord stimulation will mean there was improvement.

SECONDARY OUTCOMES:
Average Numerical Rating Scale (NRS) Pain | 2-8 days after the trial procedure
  The numeric rating scale (NRS) is a pain screening tool that uses a 0-10 scale to assess pain severity at that time, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
  Although measured at different time points, the average score for each participant is average and then summed across all participants.
Complex Regional Pain Syndrome Severity Score (CSS) | 2-8 days after the trial procedure
  A continuous score for CRPS severity. It includes 17 signs and symptoms (8 reported by the patient, 9 observed at examination date).
  A value of 50% or higher on the CSS value at postoperative follow-up (2-8 days) time point after surgery indicates success of the forward looking infrared camera.
  Although measured at different time points, the difference between the time points will be calculated and reported.
Average level of Neuropathic Pain Score (PainDetect-PD) | 2-8 days after the trial procedure
  Quantifies severity of neuropathic pain. Scores are based on patient responses to questions about pain intensity. 0 indicates no pain; 10 indicates the most pain imaginable.
  Quantitative measures (delta thermal camera value) are expected to provide a 50% or higher correlation to PD values (delta pain PD value). (The developed quantitative measurement will be compared with the currently used PD values at postoperative follow-up (2-8 days) time points after completion of the SCS.)

CONTACTS AND LOCATIONS:
Overall Officials: Semih Gungor, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: For researchers who provide a methodologically sound proposal and analyses to achieve aims in the approved proposal. Proposals should be directed to siderisa@hss.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Harden RN, McCabe CS, Goebel A, Massey M, Suvar T, Grieve S, Bruehl S. Complex Regional Pain Syndrome: Practical Diagnostic and Treatment Guidelines, 5th Edition. Pain Med. 2022 Jun 10;23(Suppl 1):S1-S53. doi: 10.1093/pm/pnac046. PMID 35687369
- [Result] Baron R, Schattschneider J, Binder A, Siebrecht D, Wasner G. Relation between sympathetic vasoconstrictor activity and pain and hyperalgesia in complex regional pain syndromes: a case-control study. Lancet. 2002 May 11;359(9318):1655-60. doi: 10.1016/S0140-6736(02)08589-6. PMID 12020526
- [Result] Croom JE, Foreman RD, Chandler MJ, Barron KW. Cutaneous vasodilation during dorsal column stimulation is mediated by dorsal roots and CGRP. Am J Physiol. 1997 Feb;272(2 Pt 2):H950-7. doi: 10.1152/ajpheart.1997.272.2.H950. PMID 9124459
- [Result] Jacobs MJ, Jorning PJ, Joshi SR, Kitslaar PJ, Slaaf DW, Reneman RS. Epidural spinal cord electrical stimulation improves microvascular blood flow in severe limb ischemia. Ann Surg. 1988 Feb;207(2):179-83. doi: 10.1097/00000658-198802000-00011. PMID 3257679
- [Result] Linderoth B, Fedorcsak I, Meyerson BA. Peripheral vasodilatation after spinal cord stimulation: animal studies of putative effector mechanisms. Neurosurgery. 1991 Feb;28(2):187-95. PMID 1671794
- [Result] Huh BK, Park CH, Ranson M, Campbell GL, Ravanbakht J. Thermogram in spinal cord stimulation with complex regional pain syndrome and a review of the literature. Neuromodulation. 2010 Apr;13(2):114-6. doi: 10.1111/j.1525-1403.2009.00236.x. Epub 2009 Sep 3. PMID 21992784
- [Result] Harden RN, Bruehl S, Stanton-Hicks M, Wilson PR. Proposed new diagnostic criteria for complex regional pain syndrome. Pain Med. 2007 May-Jun;8(4):326-31. doi: 10.1111/j.1526-4637.2006.00169.x. PMID 17610454
- [Result] Harden NR, Bruehl S, Perez RSGM, Birklein F, Marinus J, Maihofner C, Lubenow T, Buvanendran A, Mackey S, Graciosa J, Mogilevski M, Ramsden C, Schlereth T, Chont M, Vatine JJ. Development of a severity score for CRPS. Pain. 2010 Dec;151(3):870-876. doi: 10.1016/j.pain.2010.09.031. Epub 2010 Oct 20. PMID 20965657

DOCUMENTS (1):
  • Study Protocol (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT05777889/Prot_000.pdf